CLINICAL TRIAL: NCT05374447
Title: Evaluating the Diagnostic Yield and Specimen Quality With Endobronchial Ultrasound-Guided Intranodal Forceps Biopsies in Patients With Mediastinal and Hilar Lymphadenopathy: A Prospective Analysis
Brief Title: Diagnostic Yield of Intranodal Forceps Biopsies in Mediastinal Adenopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Khalil Diab, MD - Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NCR224078
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Mediastinal Lymphadenopathy; Sarcoidosis, Pulmonary; Mediastinal Diseases
Keywords: Sarcoidosis; Bronchoscopy; Endobronchial Ultrasound; Intranodal forceps biopsy
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Mediastinal Diseases; Sarcoidosis

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to EBUS-TBNA alone or EBUS-TBNA and EBUS-IFB
Who Masked: Participant
Masking Description: The participant will be blinded to which group they were randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBUS-TBNA (Active Comparator): These will be the patient who undergo EBUS-TBNA only without EBUS-IFB
  Interventions: Procedure: Endobronchial Ultrasound-Guided Intranodal Forceps Biopsy
- EBUS-TBNA + EBUS-IFB (Experimental): These will be the individuals who undergo EBUS-TBNA followed by EBUS-IFB in the same procedure
  Interventions: Procedure: Endobronchial Ultrasound-Guided Intranodal Forceps Biopsy

INTERVENTIONS:
Procedure: Endobronchial Ultrasound-Guided Intranodal Forceps Biopsy — Patients with mediastinal adenopathy will undergo EBUS-IFB and EBUS-TBNA during the same procedure to compare the yield of this procedure with EBUS-TBNA alone.
  Other Names: EBUS-IFB

SUMMARY:
The investigators will compare endobronchial ultrasound transbronchial needle aspiration (EBUS-TBNA) with intranodal forceps biopsy (EBUS-IFB) as it relates to the rate of diagnosis of suspected sarcoidosis.

DETAILED DESCRIPTION:
This is prospective, single center randomized comparative study to determine the diagnostic yield and specimen quality of endobronchial ultrasound guided intranodal forceps biopsy of patients with suspected sarcoidosis based solely on imaging. This will be a single group study and will compare transbronchial needle aspiration via 19 or 21-gauge needle with intranodal forceps biopsy.

The study aims to answer a knowledge gap a as to whether the diagnostic yield and specimen quality of EBUS-TBNA with a 19G needle is less than those obtained by 1.9mm or greater intranodal forceps biopsy. The study proposed here will add to the field by further elucidating whether this procedure is beneficial for the diagnosis as it pertains to suspected sarcoidosis.

The anticipated required enrollment is 55 patients to achieve an α of 0.05 and β of 0.2. This assumes an unassisted diagnostic yield of 62.5% with standard of care EBUS-TBNA as reported in Ray et al, and a diagnostic supplementation to 80% yield with intranodal forceps biopsies.

References

1. Oki, M., Saka, H., & Sako, C. (2004). Bronchoscopic miniforceps biopsy for mediastinal nodes. Journal of Bronchology & Interventional Pulmonology, 11(3), 150-153.
2. Herth FJ, Morgan RK, Eberhardt R, Ernst A. Endobronchial ultrasound-guided miniforceps biopsy in the biopsy of subcarinal masses in patients with low likelihood of non-small cell lung cancer. Ann Thorac Surg. 2008 Jun; 85(6):1874-8.
3. Chrissian A, Misselhorn D, Chen A. Endobronchial-ultrasound guided miniforceps biopsy of mediastinal and hilar lesions. The Annals of Thoracic Surgery. 2011;92(1):284-288.
4. Franke KJ, Bruckner C, Szyrach M, Ruhle KH, Nilius G, Theegarten D. The contribution of endobronchial ultrasound-guided forceps biopsy in the diagnostic workup of unexplained mediastinal and hilar lymphadenopathy. Lung. 2012;190(2):227-232.
5. Herth FJF, Schuler H, Gompelmann D, et al. Endobronchial ultrasound-guided lymph node biopsy with transbronchial needle forceps: a pilot study. European Respiratory Journal. 2012;39(2):373-377.
6. Darwiche K, Freitag L, Nair A, et al. Evaluation of a novel endobronchial ultrasound-guided lymph node forceps in enlarged mediastinal lymph nodes. Respiration. 2013;86(3):229-236.
7. Ray AS, Li C, Murphy TE, et al. Improved diagnostic yield and specimen quality with endobronchial ultrasound-guided forceps biopsies: a retrospective analysis. The Annals of Thoracic Surgery. 2020;109(3):894-901

ELIGIBILITY:
Inclusion Criteria:

* Radiologic evidence of mediastinal and/or hilar lymphadenopathy
* Attending radiologist or pulmonologist reports a possible diagnosis of sarcoidosis
* Age 18 years or older

Exclusion Criteria*:

These are the characteristics that a participant must NOT have in order to be eligible to participate in the study.

Order Number Criteria

* Severe pulmonary hypertension
* Inability to undergo general anesthesia
* Severe coagulopathy or bleeding diathesis
* Previously diagnosed sarcoidosis
* Patient presently taking clopidogrel
* Patient deemed to be high risk for general anesthesia per anesthesiologist
* Hemodynamic instability
* Mediastinitis
* Acute Hypercarbic Respiratory Failure (pCO2 >55mmHg)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield | 1 year
  Diagnostic yield of EBUS-TBNA + EBUS-IFB compared to EBUS-TBNA alone

SECONDARY OUTCOMES:
Duration of Procedure | 1 year
  Duration of combined EBUS-TBNA +IFB procedure compared to TBNA alone
Complications | 1 year
  Complications of EBUS-TBNA +IFB procedure compared to TBNA alone

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Gomberg, MD, Study Director — The George Washington University
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No